CLINICAL TRIAL: NCT04659356
Title: Evaluation of a SARS-CoV-2 Infectious Risk Management Protocol on the Transmission of Nosocomial COVID in Intensive Care Unit"
Brief Title: NOSOcomial COVID-19 in ICU (NOSOCOVID)
Acronym: NOSOCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR_NOSOCOVID
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infectious Disease (COVID-19); Nosocomial Infection; Nosocomial COVID-19
Keywords: Coronavirus Infectious Disease (COVID-19); Nosocomial Infection; SARS-Coronavirus-2; Intensive Care Units (ICU); Personal protective equipment
MeSH Terms: conditions — COVID-19; Cross Infection | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted in Intensive Care Units: All patients admitted in our ICU since august were enrolled in our study, after they have been informed and given their consent for their participation in this observational study.
  Interventions: Other: Patients admitted in Intensive Care Units

INTERVENTIONS:
Other: Patients admitted in Intensive Care Units — Data will be collected computerized patient records by the clinicians in charge of the patient.

SUMMARY:
The current global pandemic at COVID-19 is a major public health issue. Transmission of the virus is primarily through direct and close person-to-person contact. The protection of health care personnel and the limitation of transmission of nosocomial COVID is paramount. Protective measures have already shown their effectiveness in limiting the spread of the virus: the use of masks, the wearing of protective gowns, the wearing of protective eyewear, social and physical distancing. A recent U.S. study (Rhee et al. JAMA 2020) reported a very low incidence of 1.7% of nosocomial COVID, but this was achieved with the application of rigorous infection risk management protocols. In addition to the widespread use of masks and protective measures, dedicated COVID units had been created, with air treatment. The implementation of these dedicated units requires the mobilization of considerable human and material resources, which is not feasible in all hospitals over the long term.

In view of the second wave of the epidemic in France, with the rising numbers of new cases of COVDI-19 admitted to intensive care units since the end of the summer 2020, it is essential to organize the intensive care units to ensure the protection of personnel and limit the risk of nosocomial COVID-19, while continuing to care for non-COVID patients.

In Intensive Care unit (ICU) at the Nantes University Hospital, a strict protocol for the management of suspected or confirmed COVID patients has been in place since early september 2020. The objective of this study is to evaluate the effectiveness of this protocol for managing the infectious risk of SARS-COV-2 on the incidence of nosocomial COVID in patients admitted in ICU. The secondary objectives are to evaluate the incidence of nosocomial-associated COVIDs contracted by caregivers, and the incidence of asymptomatic positive SARS-CoV-2 cases in ICU.

DETAILED DESCRIPTION:
All patients admitted in our ICU since august 2020 were enrolled in the study, after they have been informed and given their consent for their participation in this observational study. Data will be collected computerized patient records by the clinicians in charge of the patient.

Because of variants emergence, the investigators decided to had a second period from march to july. The investigators anticipate an inclusion of approximately 1000 patients.

In an observational study, there is no risk to the patient

ELIGIBILITY:
Inclusion Criteria:

* All Patients admitted in ICU during the inclusion period (Nantes University Hospital)
* AND all Healthcare workers working in ICU during the inclusion period (Nantes University Hospital)

Exclusion Criteria:

* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU and Healthcare workers working in ICU
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of nosocomial COVID-19 | up to 10 months
  Occurence of a nosocomial COVID-19 that is certain or probable. Community-acquired certain and probable COVIDs will be excluded from the main analysis.
  The incidence rate of nosocomial COVID will be expressed in patient-days:
  Ratio of the number of patients with nosocomial COVID to the sum of exposure times, i.e. :
  * for patients without nosocomial COVID: duration of hospitalization in ICU
  * for patients presenting with nosocomial COVID: delay between the date of the start of hospitalization in ICU and the occurrence of nosocomial COVID.

SECONDARY OUTCOMES:
Occurrence of a nosocomial COVID-19 that is certain and Occurrence of a nosocomial COVID-19 that is probable. | up to 10 months
  Prevalence of community-acquired COVID that is certain and Prevalence of community-acquired COVID that is probable.
  Prevalence of nosocomial and community-acquired COVID in healthcare workers. Prevalence will be defined as the ratio of the number of caregivers developing a COVID to the number of caregivers working in ICU during the inclusion period.
  Prevalence of patients with SARS-CoV-2 positive samples but asymptomatic in ICU.
  Risk factors to development a nosocomial COVID (certain and probable).
evaluate the occurence | up to 12 months
  * ICU nosocomial infections rates (ventilator associated acquired pneumonia)
  * Highly resistant bacteria colonization and infection acquired in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France